CLINICAL TRIAL: NCT07389668
Title: The Effect of the Use of Hand Massage Stimulation Techniques on the Severity of Nausea-Vomiting and Quality of Life in Pregnant Women Diagnosed With Hyperemesis Gravidarum
Brief Title: The Effect of the Use of Hand Massage Stimulation Techniques on the Hyperemesis Gravidarum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra Nur Emre, PhD student, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/128
Record Dates: First submitted 2026-01-27; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy Related
Keywords: Nausea-vomiting; quality of life; pregnancy; massage; midwife

STUDY DESIGN:
Intervention Model Description: randomized controlled trial conducted with experimental and control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard maintenance (No Intervention): Group not receiving seed therapy (su jok)
- seed therapy (su jok) (Experimental): Group that received seed therapy (su jok)
  Interventions: Other: seed therapy (su jok)

INTERVENTIONS:
Other: seed therapy (su jok) — In hand massage, tiny swellings called "ball conformity" occur on the reflection points of the organs where the complaint occurs on the hands and feet. It is argued that the sensitivity of the relevant point to pressure has a direct correlation with the level of pain in the body part. A rod called a "diagnostic probe" or "diagnostic rod" made of metal, plastic or wood, approximately ten centimeters long, is used to detect the painful point on the hand and foot. After the correct point is detected, various techniques are applied to stimulate these points and ensure the continuation of the energy flow.In this study, the seed massage technique, which does not cause any side effects among the hand massage stimulation methods, requires a basic level certificate for its use, does not require being a health professional, and can be easily applied by anyone, will be used. Seed massage is a method applied by first detecting pain through a probe on the points of the organs reflected on the hand
  Arms: seed therapy (su jok)

SUMMARY:
The aim of this study is to determine the effect of the use of hand massage stimulation techniques on nausea-vomiting severity and quality of life in pregnant women diagnosed with hyperemesis gravidarum.

Research Hypotheses H1-a: The use of hand massage stimulation techniques in pregnant women diagnosed with hyperemesis gravidarum reduces the severity of nausea-vomiting.

H1-b: The use of hand massage stimulation techniques in pregnant women diagnosed with hyperemesis gravidarum increases the quality of life.

Data will be collected from pregnant women diagnosed with hyperemesis gravidarum in the maternity ward. It will be ensured that the midwifery intervention is implemented in a way that does not disrupt the examination routine. Seed therapy (su-jok) will be applied by researcher Esra Nur Emre, who has a basic level su jok therapy certificate.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of the use of hand massage stimulation techniques on nausea-vomiting severity and quality of life in pregnant women diagnosed with hyperemesis gravidarum.

Data will be collected from pregnant women diagnosed with hyperemesis gravidarum in the maternity ward of Hatay Dörtyol State Hospital. Participants who meet the inclusion criteria and agree to participate will be informed about the study and participants who fill out the "Minimum Informed Consent Form" will be included in the study. Data collection tools will be applied to pregnant women who agree to participate in the study by the researcher through face-to-face interviews. Data collection forms will be applied by the researcher, paying attention to patient privacy, and the pre-test data collection phase will be completed. After the pre-test data collection phase is completed, hand stimulation techniques (su-jok seed therapy) will be applied to the pregnant women in the experimental group by the researcher. After the pregnant women are given detailed information about the application, pain points will be determined according to the organ reflections on the hand. Green mung bean seeds, which are seeds used for nausea, will be fixed on the detected points and the fixed seed will be removed after 5-6 hours. The experimental group will be completed in two sessions in 24 hours. The second session will start with correct point detection and proceed in the same way as the first session. The procedure will be terminated after 5-6 hours. The PUQE (Nausea and Vomiting Severity Evaluation in Pregnancy) Test and the SF 36 Quality of Life Scale will be re-applied from the data collection forms. No intervention will be applied to the women in the control group, however, the Personal Information Form, Visual Analog Scale, PUQE (Nausea and Vomiting Severity Evaluation in Pregnancy) Test and the SF 36 Quality of Life Scale will be applied simultaneously with the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are over 18 years old,
* Who can read and write,
* Who do not have any psychiatric disorders,
* Who are not experiencing a risky pregnancy,
* Who are hospitalized with a diagnosis of hyperemesis gravidarum,
* Who do not react negatively to any interventions aimed at touch, such as massage,
* Who have full and healthy tissue integrity in the area where the massage will be performed

Exclusion Criteria:

* Those whose pregnancy has ended for any reason,
* Those who have not been hospitalized despite being diagnosed,
* Pregnant women in the third trimester of pregnancy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Nausea-vomiting severity scores | Data collection forms were administered by the researcher using face-to-face interviews in the first stage (days 1-2 and 3), telephone interviews in the second stage (day 15), and face-to-face interviews again in the third stage (days 30-31).
  The Pregnancy Nausea and Vomiting Severity Assessment Test (PUQE) is a scoring system used to measure the severity of nausea and vomiting during pregnancy. The lowest score on the scale is 3 and the highest is 15. 0-3 indicates no symptoms, 4-6 indicates mild, 7-12 indicates moderate and 13-15 indicates severe nausea and vomiting during pregnancy.

SECONDARY OUTCOMES:
Quality of life scores | Data collection forms were administered by the researcher using face-to-face interviews in the first stage (days 1-2 and 3), telephone interviews in the second stage (day 15), and face-to-face interviews again in the third stage (days 30-31) .
  SF-36 quality of life scale includes SF-36 YKÖ sub-dimensions of physical function 3rd question (options a, b, c, d, e, f, g, h, ı, j), social function 6th and 10th questions, physical role difficulty 4th question (options a, b, c, d), emotional role difficulty 5th question (options a, b, c), mental health 9th question b, c, d, f, h options, vitality/energy 9th question a, e, g, i options, pain 7th and 8th questions, general health 1st, 2nd and 11th questions (options a, b, c, d). SF-36 YKÖ is scored in a way that as the scores in the sub-dimensions increase, the quality of life also increases. With SF-36 YKÖ, both comprehensive quality of life and all sub-dimensions of quality of life are evaluated. The total score is between 0-100. As a result, a score of 0 indicates the worst health status, and a score of 100 indicates the best health status.

CONTACTS AND LOCATIONS:
Overall Officials: Esra GÜNEY, PhD, Principal Investigator — İnonu Üniversity
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research results will be shared.

REFERENCES:
- See also: Reference Link — https://pubmed.ncbi.nlm.nih.gov/19879515/